CLINICAL TRIAL: NCT02001649
Title: Genetic Variants Associated With Adolescent Suicide Attempts: a Candidate-gene Association Study.
Brief Title: Genetic Variants Associated With Adolescent Suicide Attempts
Acronym: VGTSA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Rouen (Other)
Collaborators: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: 2013/092/HP
Record Dates: First submitted 2013-11-14; First posted 2013-12-05 (Estimated); Last update posted 2016-10-10 (Estimated); Status verified 2016-10

CONDITIONS: Attempt Suicide
Keywords: suicide; adolescent; genetic; SNP
MeSH Terms: conditions — Suicide, Attempted; Suicide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Inpatient group SNP Genotyping (Other): Patients will be recruited from pediatric departments in which 13 -17 y old adolescents are hospitalized for a suicide attempt. Data will be collected through self-administered questionnaires and face to face interview. DNA will be extracted from saliva sample.
  Individuals will be genotyped at a total of 96 SNPs
  Interventions: Genetic: SNP Genotyping
- Control group SNP Genotyping (Other): Control subjects are young adults without suicide attempt and without mental disorders
  Interventions: Genetic: SNP genotyping

INTERVENTIONS:
Genetic: SNP Genotyping — Individuals were genotyped at a total 96 SNP from 15 candidate gene
  Arms: Inpatient group SNP Genotyping
Genetic: SNP genotyping
  Arms: Control group SNP Genotyping

SUMMARY:
Suicidal behaviors is known to aggregate in families. The purpose of this study is to evaluate association between common polymorphisms in genes important for neurobiological pathways linked to suicidal behaviors and suicide attempt among adolescents patient.

DETAILED DESCRIPTION:
In France, suicide is the second leading cause of death among the 14-22 years population. Suicide behavior (SB) spans a spectrum ranging from suicidal ideation to suicide attempts and completed suicide. Several factors likely determine the predisposition to SB, including biological factors and psychosocial stressors. For biological factors, convergent evidence from adoption, family, and twin studies of suicide strongly suggests genetic contributions to liability for SB. Although genetic factors play a role in SB, identifying specific genes involved has proved challenging. Molecular-genetic technologies have made great advances in the past decade, including genome- wide searches for disease-causing genes with the linkage disequilibrium (LD) approach. Despite being a major public health problem in the youth population, genetic associations studies regarding suicidal behavior in adolescence are still rare. Genes that code for proteins involved in regulating serotonergic neurotransmission have thus been major candidate genes for association studies of SB. Among them, genes for serotonin metabolism (tryptophan hydroxylase, TPH), serotonin transport (5-HTT), and the serotonergic 2A (5-HT2A) receptor have received the most research attention.

The identification of relevant genetic variants or SNPs in others genes which are involved in the neurobiological pathways (which the alteration may contribute to a suicidal behavior) can help not only to advance knowledge of the genetic bases of suicide but also to identify new therapeutic targets.

On the basis of review of the literature, investigators will identify candidate genes that have been reported to be associated with suicidal events.

The investigators will target genes related to central serotonergic and noradrenergic neurotransmission, and monoamine metabolism (MAOA). The investigators will also study genes involved in glutamatergic neurotransmission (GRIK2, GRIA3) and in the HPA axis (FKBP5) and genes that code for neurotrophic proteins (BDNF).

DNA will be obtained from saliva. All genotyping will be carried out using standard polymerase chain reaction-based techniques that are routinely used in the Human Genetics Laboratory. DNA segments containing the target variable site will be amplified using unique sequence flanking primers.

Tests of association between genetic variant and suicide attempt will be conducted using Chi squared and Armitage Trend Tests. Logistical regression analyses will be performed to evaluate the contribution of individual genetic variant to the prediction of suicide attempt, and to examine SNPs for potential gene-gene and gene-environment interactions.

ELIGIBILITY:
Inclusion Criteria:

Case :

* Age at admission between 13 and 17 years old
* Hospitalized for attempted suicide
* Absence of prominent mental retardation or organic brain damage
* Fluent in French
* Able to comprehend the study procedures and to undergo entry assessments safely
* Provided written informed consent for study participation, and additional consent from the patient's parents or guardians
* Northern and Western European ancestry (HapMap-CEU)
* Medical insurance coverage

Control :

* Healthy adult volunteers
* No present or past psychiatric illness
* No personal history of suicidal behavior and without a family history of suicide
* Provided written informed consent for study participation
* Northern or Western European ancestry (HapMap-CEU)
* Medical insurance coverage

Exclusion Criteria:

Case:

* Inability to get an informed and valid consent
* Home address outside the selected hospitals' geographic areas
* Intellectual disability or organic brain damage
* Origine ethnique non CEU
* Absence of medical insurance coverage
* Pregnant or lactating women
* Without Northern or Western European ancestry (HapMap-CEU)

Control :

* Inability to get an informed and valid consent
* Intellectual disability or organic brain damage
* History of suicidal behavior
* Psychiatric disorder, past or present
* Family history of suicide
* Borderline personality disorder
* Absence of medical insurance coverage
* Pregnant or lactating women
* Without Northern or Western European ancestry (HapMap-CEU)

Ages: 13 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 250 (Actual)
Dates: Start 2013-12; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Odds ratio (OR) and 95% confidence interval (CI) will be estimated using a logistic regression model to assessing the contribution of each polymorphism as a risk factor in predicting suicidal behavior | Between day 1 and day 5 during hospitalization
  Measure is a composite outcome measure consisting of multiple measures
  Post hoc Bonferroni correction will be employed to correct for multiple testing.
  Chi- square test will performed to analyze genetic associations

CONTACTS AND LOCATIONS:
Overall Officials: BOJAN MIRKOVIC, MD, Principal Investigator — CHU Rouen, Fédération de pédopsychiatrie du Pr Gérardin
Locations (1):
- Chu Rouen, Rouen, Haute Normandie, France